CLINICAL TRIAL: NCT05644990
Title: Direct Detection of ESKAPE Pathogens From Whole Blood Using T2MR Bacteria Panel in Patients With Pyogenic Spondylodiscitis and Infective Endocarditis
Brief Title: T2MR PCR Detection of ESKAPE Pathogens in Patients With Pyogenic Spondylodiscitis and Infective Endocarditis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Bulovka Hospital (Other); University Hospital, Motol (Other)
Responsible Party: Sponsor
Other Study IDs: 22-IGS06-36
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2022-12

CONDITIONS: Osteomyelitis; Vertebra; Endocarditis, Bacterial
Keywords: Spondylodiscitis; Endocarditis; PCR; T2Bacteria Panel; MRI
MeSH Terms: conditions — Osteomyelitis; Endocarditis, Bacterial; Discitis; Endocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — 4 ml whole blood sample drawn into the K2EDTA vacutainer (BD367861/BD367862/BD368861)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T2Bacteria Panel positive: Patients with spondylodiscitis and endocarditis who had positive T2Bacteria Panel test.

SUMMARY:
Our prospective observational study focuses on the rapid detection of etiologic agents of pyogenic spondylodiscitis and infective endocarditis using the T2 Bacteria Panel (T2Biosystems). This diagnostic method combines polymerase chain reaction (PCR) and T2 magnetic resonance for detection of bacterial DNA from whole blood samples. It detects six pathogens known by the acronym ESKAPE (E. coli, S. aureus, K. pneumoniae, A. baumannii, P. aeruginosa, and E. faecium). In recent years, similar studies using the Bacteria Panel and Candida Panel have been performed in patients with bloodstream infections, leaving us with optimistic results.The aim of this study is to verify whether T2B can identify the etiologic agents of localized infections, specifically spondylodiscitis and endocarditis, with better sensitivity and specificity and shorter time to result compared to conventional diagnostics from blood culture. Rapid detection of pathogen may reduce time to targeted pathogen-specific antibiotic therapy and subsequently improve outcomes, shorten the treatment and contribute to slowing the development of antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spondylodiscitis or/and facet joint infection or/and sacroileitis
* Diagnosis of infective endocarditis
* Antibiotic treatment not received or not longer than 24 hours
* Ability to give informed consent

Exclusion Criteria:

* Spine infection or/and endocarditis not confirmed
* Antibiotic treatment longer than 24 hours
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with pyogenic spine infections and/or infective endocarditis, treated at the standard care wards and ICU of the Department of infectious diseases and Department of orthopaedics of the University Hospital Bulovka.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the T2 Bacteria Panel | 3 years
  Sensitivity and specificity of the T2 Bacteria Panel for ESKAPE pathogens direct detection in patients investigated for suspected pyogenic vertebral infection and/or infective endocarditis, compared with conventional blood culture and/or other relevant biological samples culture .
Expected treatment outcomes in patients diagnosed by T2 Bacteria Panel | 4 years
  T2 Bacteria Panel is expected to shorten the time to result compared to conventional methods. Rapid detection of the bacteria followed by early pathogen-specific antibiotic therapy should improve the outcomes of patients with spondylodiscitis and infective endocarditis, e.g. mortality, morbidity and length of treatment.

SECONDARY OUTCOMES:
Diagnostic utility of T2 Bacteria Panel in other localized infections | 4 years
  Patients with other localized infections (other than spine or endocardium infections) who were tested with T2 Bacteria Panel before their diagnosis was assessed, will be excluded from the study. They will be separately evaluated to find out if T2MR diagnostics is useful also in other localised infections (besides of spine infection and endocarditis).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bulovka, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No